CLINICAL TRIAL: NCT02527421
Title: A Randomized, Parallel Group, Open-Label, Multicenter Study to Assess the Potential for Adrenal Suppression and Systemic Drug Absorption Following Multiple Dosing With DFD-01 (Betamethasone Dipropionate) Spray, 0.05%
Brief Title: DFD01 Spray HPA Axis Suppression Study in Adolescent Patients With Moderate to Severe Plaque Psoriasis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Not able to recruit patients with the current enrollment criteria.
Sponsor: Primus Pharmaceuticals (Industry)
Collaborators: Prosoft Clinical (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DFD01-CD-013
Record Dates: First submitted 2015-08-10; First posted 2015-08-19 (Estimated); Results first posted 2021-10-21 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Plaque Psoriasis
MeSH Terms: interventions — Betamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DFD01 Spray Group 1 (Experimental): DFD01 spray, twice daily, 15 days
  Interventions: Drug: DFD01 Spray
- DFD01 Spray Group 2 (Experimental): DFD01 spray, twice daily, 29 days
  Interventions: Drug: DFD01 Spray

INTERVENTIONS:
Drug: DFD01 Spray — DFD-01 (betamethasone dipropionate) Spray, 0.05%
  Other Names: betamethasone

SUMMARY:
To evaluate the potential of DFD-01 (betamethasone dipropionate) Spray, 0.05% to suppress the hypothalamic-pituitary-adrenal (HPA) axis.

DETAILED DESCRIPTION:
To evaluate the potential of DFD-01 (betamethasone dipropionate) Spray, 0.05% to suppress the hypothalamic-pituitary-adrenal (HPA) axis when applied twice daily for 15 days or when applied twice daily for 29 days, in adolescent subjects with moderate to severe plaque psoriasis under maximal use conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must weigh at least 55 pounds
2. Subjects must present with a clinical diagnosis of stable (at least 3 months) plaque psoriasis.
3. Subjects with psoriasis involving ≥ 10% BSA, not including the face, scalp, groin, axillae and other intertriginous areas..
4. Subjects must have moderate to severe plaque psoriasis at the Baseline Visit.
5. Subjects whose results from the screening ACTH stimulation test are considered normal (cortisol level >18 ug/dL at 30 minutes post stimulation) and show no other signs of abnormal HPA axis function or adrenal response.

Exclusion Criteria:

1. Current diagnosis of unstable forms of psoriasis including guttate, erythrodermic, exfoliative or pustular psoriasis.
2. History of organ transplant requiring immunosuppression, HIV, or other immunocompromised state.
3. Have received treatment for any type of cancer within 5 years of the Baseline Visit.
4. Use within 60 days prior to the Baseline Visit of: 1) immunosuppressive drugs (e.g., tacrolimus, pimecrolimus), 2) systemic antipsoriatic treatment (e.g., methotrexate, cyclosporine, hydroxyurea), or 3) biologic treatment for psoriasis (e.g., infliximab, adalimumab, etanercept, ustekinumab, secukinumab, or alefacept).
5. Use within 30 days prior to the Baseline Visit of: 1) topical antipsoriatic drugs (salicylic acid, anthralin, coal tar, calcipotriene), 2) PUVA therapy, 3) systemic anti-inflammatory agents (e.g., mycophenolate mofetil, sulfasalazine, 6-thioguanine), or 4) UVB therapy.
6. Use within 30 days prior to the Screening Visit of any product containing corticosteroids. Inhaled, intraocular, intranasal, etc. steroids are not allowed.
7. Subjects who have an abnormal sleep schedule or work overnight.
8. Subjects with a known history of acute adrenal crisis, Addison's disease or decreased adrenal output, low pituitary function or pituitary tumors.
9. Subjects who have a history of an adverse reaction to cosyntropin injection or similar test reagents.

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3 (Actual)
Dates: Start 2015-08-19 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Srinivas Sidgiddi, MD, Study Director — Dr. Reddy's Laboratories, Inc
Locations (8):
- United States (8):
  - Site 102, Encino, California
  - Site 104, Irvine, California
  - Site 100, San Diego, California
  - Site 109, Lebanon, New Hampshire
  - Site 107, New York, New York
  - Site 106, Arlington, Texas
  - Site 101, Houston, Texas
  - Site 105, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | DFD01 Spray Group 1 | DFD01 Spray Group 2
Started | 2 | 1
Completed | 1 | 1
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DFD01 Spray Group 1 | DFD01 Spray Group 2 | Total
Number analyzed (Participants) | 2 | 1 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 1 | 3
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Participants With HPA Axis Suppression at End of Treatment (Day 15 or Day 28) With Recovery 29 Days Later
Description: Number of participants with HPA axis suppression at End of Treatment (day 15 or day 28) with recovery 29 days later, by measuring the level of cortisol in the blood after ACTH stimulation test
Time Frame: End of Treatment (day 15 or day 28) with recovery 29 days later
Population: Subjects who completed the treatment period
Measure: Count of Participants; unit: Participants
Arm/Group | DFD01 Spray Group 1 | DFD01 Spray Group 2
Number analyzed (Participants) | 1 | 1
Participants | 0 | 1

2. Primary Outcome: Participants With HPA Axis Suppression at Day 29
Description: Number of participants with HPA axis suppression at Day 29, by measuring the level of cortisol in the blood after ACTH stimulation test
Time Frame: Day 29
Measure: Count of Participants; unit: Participants
Arm/Group | DFD01 Spray Group 1 | DFD01 Spray Group 2
Number analyzed (Participants) | 1 | 1
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: 43 days (14-day treatment group) or 57 days (29-day treatment group)
Arm/Group | DFD01 Spray Group 1 | DFD01 Spray Group 2
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 1/2 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DFD01 Spray Group 1 (N=2) | DFD01 Spray Group 2 (N=1)
HPA Axis suppression (Endocrine disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No report, abstract, oral presentation, or publication of the results of the Study proposed by Institution shall be presented or published without the prior written consent of the Sponsor or as otherwise permitted for regulatory agency inspections.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-13): https://cdn.clinicaltrials.gov/large-docs/21/NCT02527421/Prot_SAP_000.pdf